CLINICAL TRIAL: NCT03821584
Title: Brain Perfusion Assessment in the Acute Phase of Migraine Aura.
Acronym: PERCAM
Status: Terminated | Type: Observational
Why Stopped: Recruiting terminated
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC18_0373
Record Dates: First submitted 2019-01-04; First posted 2019-01-30 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-07

CONDITIONS: Emergencies
Keywords: migraine; perfusion arterial; aura brain
MeSH Terms: conditions — Emergencies; Migraine Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: the difference of care management and prognosis, an early distinction of migraine aura based on imaging techniques will have a particular interest — the difference of care management and prognosis, an early distinction of migraine aura based on imaging techniques will have a particular interest

SUMMARY:
The aim of the study is to determine the proportion of patients with change in brain perfusion during the acute phase of migraine attack with aura.

DETAILED DESCRIPTION:
Migraine is a benign and frequent disorder. Migraine aura consists in reversible focal neurological symptoms developing gradually during attack. Its diagnosis relies mainly on patient's history, clinical examination and exclusion of other possible secondary causes to explain transient neurological signs. Thus it can be difficult particularly during first attack or during attack without headache to differentiate migraine aura from transient ischemic stroke. Considering the difference of care management and prognosis, an early distinction of migraine aura based on imaging techniques will have a particular interest. MRI with diffusion, SWI, Flair 2D, ARM 3D TOF, ASL sequences' are routinely performed for the management of acute neurological deficit. Arterial spin labeling (ASL), as a MR perfusion method, will be used to describe brain perfusion during migraine aura. The study hypothesis is that hyperperfusion occurs in brain territories corresponding to the neurological symptoms during migraine aura.

ELIGIBILITY:
Inclusion Criteria:

* Age between greater than or equal to 18
* Able to undergo MRI during migraine aura

Exclusion Criteria:

* Pregnant females
* Contraindications towards MRI scanning
* History of epilepsy, psychiatric disease, or any other neurologic disease (brain tumors, stroke..).
* Presence of abnormalities on the MRI that could explain the neurological deficit.
* Adults under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital with neurological deficit and final clinical diagnosis of migraine with aura (certain probable as defined by The International Classification of Headache Disorders)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Perfusion pattern of concerned brain areas | 1 hour
  Presence or absence of hypo-hyperperfusion using arterial spin labeling. Visual assessments and comparison between hemispheres

SECONDARY OUTCOMES:
Pattern of perfusion and aura duration | 12 month
  Change in brain perfusion in relation to neurological deficits (migraine aura) duration.

CONTACTS AND LOCATIONS:
Overall Officials: Solene de Gaalon, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU Nantes, Nantes, France